CLINICAL TRIAL: NCT05687955
Title: Exercise Rehabilitation for Hip-related Pain and Dysfunction in Full Time Student Circus Arts Performers: a Pilot Trial
Brief Title: Exercise Rehabilitation for Hip-related Pain and Dysfunction in Student Circus Arts Performers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swinburne University of Technology (Other)
Collaborators: National Institute of Circus Arts (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SwinburneUT
Record Dates: First submitted 2023-01-04; First posted 2023-01-18 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Hip Dysplasia; Femoro Acetabular Impingement
MeSH Terms: conditions — Hip Dislocation; Femoracetabular Impingement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hip Exercise Program (Experimental): A 12-week strength exercise protocol has been specifically designed to focus on hip rehabilitation appropriate for circus performance.
  Interventions: Other: Hip Exercise Program

INTERVENTIONS:
Other: Hip Exercise Program — The exercise intervention is being implemented 3 times per week. Two sessions can be completed at home by the participant, and one session per week will be attended by a physiotherapist that will monitor exercise technique and progress the exercise program for each participant. The exercise protocol has been specifically designed to focus on hip rehabilitation appropriate for circus performance. The exercise program will involve hip strength exercises in the sagittal, coronal and transverse planes using weights and elastic bands (Theraband). It will also include trunk strength and postural correction exercises to address swayback posture which is a common clinical presentation in those with hip dysplasia.

SUMMARY:
Hip injuries are reported to account for 71% and 29% of all injuries reported in female and male performers, respectively, at the National Institute of Circus Arts. There are no reports on hip pathology in circus performers, nor are there any reported exercise interventions for hip pain in circus performers.

This study aims to:

To assess the effect of an exercise rehabilitation program on patient-reported outcome measures, hip strength and range of movement, and functional assessments in circus arts students with clinically and radiologically diagnosed hip pain-related disorders.

Participants will undertake a 12-week strength exercise protocol that has been specifically designed to focus on hip rehabilitation appropriate for circus performance. Expected outcome: Improvements in patient reported outcome measure (PROM) scores and an increase in function, strength and hip range of movement in people with hip pain

ELIGIBILITY:
Inclusion Criteria:

* 3-month history hip/groin pain +/- symptoms including clicking, giving way, locking, or catching, one or more of a positive
* positive FADIR pain provocation test
* positive HEER test (hip extension and external rotation)
* positive prone instability test
* imaging to support a pathological hip (e.g., CAM morphology, hip dysplasia)

Exclusion Criteria:

* OA degree >1 on classification of Tönnis
* Centre Edge-angle <10 degrees
* Legg-Calvé-Perthes or epiphysiolysis
* history of hip joint surgery or significant hip trauma (fracture +/- dislocation)
* neurologic motor deficit (lower limb power, strength or reflex deficit)
* hip pain from a lumbar origin (positive passive straight leg raise, combined lumbar extension and rotation)
* connective tissue disorder (e.g., Ehlers-danlos or Marfan syndrome)
* pregnancy or breastfeeding.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
The Copenhagen Hip and Groin Outcome Score (HAGOS) | Baseline
  Patient Reported Outcome Measure, score on 0-100 scale, with zero representing extreme hip and/or groin problems and 100 representing no hip and/or groin problems.
The Copenhagen Hip and Groin Outcome Score (HAGOS) | 3-months
  Patient Reported Outcome Measure, score on 0-100 scale, with zero representing extreme hip and/or groin problems and 100 representing no hip and/or groin problems.
The Copenhagen Hip and Groin Outcome Score (HAGOS) | 6-months
  Patient Reported Outcome Measure, score on 0-100 scale, with zero representing extreme hip and/or groin problems and 100 representing no hip and/or groin problems.
The Copenhagen Hip and Groin Outcome Score (HAGOS) | 9-months
  Patient Reported Outcome Measure, score on 0-100 scale, with zero representing extreme hip and/or groin problems and 100 representing no hip and/or groin problems.
International Hip Outcome Tool (iHOT-12) | Baseline
  Patient Reported Outcome Measure, scored using a visual analog scale from 0 to 100, with a score of 100 being the best function and least amount of symptoms
International Hip Outcome Tool (iHOT-12) | 3-months
  Patient Reported Outcome Measure scored using a visual analog scale from 0 to 100, with a score of 100 being the best function and least amount of symptoms
International Hip Outcome Tool (iHOT-12) | 6-months
  Patient Reported Outcome Measure scored using a visual analog scale from 0 to 100, with a score of 100 being the best function and least amount of symptoms
International Hip Outcome Tool (iHOT-12) | 9-months
  Patient Reported Outcome Measure scored using a visual analog scale from 0 to 100, with a score of 100 being the best function and least amount of symptoms
European Quality of life questionnaire (EQ-5D-5L) | Baseline
  Patient Reported Outcome Measure
European Quality of life questionnaire (EQ-5D-5L) | 3-months
  Patient Reported Outcome Measure
European Quality of life questionnaire (EQ-5D-5L) | 6-months
  Patient Reported Outcome Measure
European Quality of life questionnaire (EQ-5D-5L) | 9-months
  Patient Reported Outcome Measure
Tampa Scale of Kinesiophobia (TSK) | Baseline
  Patient Reported Outcome Measure
Tampa Scale of Kinesiophobia (TSK) | 3-months
  Patient Reported Outcome Measure
Tampa Scale of Kinesiophobia (TSK) | 6-months
  Patient Reported Outcome Measure
Tampa Scale of Kinesiophobia (TSK) | 9-months
  Patient Reported Outcome Measure
Hip Strength assessment | Baseline
  Strength of hip abduction, adduction, sitting hip flexion at 90deg, prone extension with knee extended, prone external and internal rotation will be measured using a hand-held dynamometer.
Hip Strength assessment | 9-months
  Strength of hip abduction, adduction, sitting hip flexion at 90deg, prone extension with knee extended, prone external and internal rotation will be measured using a hand-held dynamometer.
Hip Range of Motion | Baseline
  Hip flexion, Hip internal rotation and external rotation will be measured using an inclinometer
Hip Range of Motion | 9-months
  Hip flexion, Hip internal rotation and external rotation will be measured using an inclinometer

SECONDARY OUTCOMES:
Functional movement screen Y-balance test | Baseline
  This will measure a circus performers capacity to stand on one leg and reach their opposite leg as far as possible forwards, backwards and sideways. This provides a measure of both strength and flexibility, has been used in prior hip research, and shown to have excellent intra and inter-rater reliability.
Functional movement screen Y-balance test | 9-months
  This will measure a circus performers capacity to stand on one leg and reach their opposite leg as far as possible forwards, backwards and sideways. This provides a measure of both strength and flexibility, has been used in prior hip research, and shown to have excellent intra and inter-rater reliability.
Single leg Hop for distance | Baseline
  The distance of a participant hop will be measured, taking off and landing on the same foot, maintaining their balance for about 2-3 seconds on landing. The best of three hops will be recorded.
Single leg Hop for distance | 9-months
  The distance of a participant hop will be measured, taking off and landing on the same foot, maintaining their balance for about 2-3 seconds on landing. The best of three hops will be recorded.
Trunk Muscle Endurance Test | Baseline
  The duration of a side-plank will be recorded in seconds/minutes. The test will be ceased after 3 minutes.
Trunk Muscle Endurance Test | 9-months
  The duration of a side-plank will be recorded in seconds/minutes. The test will be ceased after 3 minutes.
One leg rise test | Baseline
  The number of sit to stand movements on a single leg performed from a starting position where the knee is at 90deg will be recorded. The test will be ceased if the participant reaches 50 one leg rises.
One leg rise test | 9-months
  The number of sit to stand movements on a single leg performed from a starting position where the knee is at 90deg will be recorded. The test will be ceased if the participant reaches 50 one leg rises.

CONTACTS AND LOCATIONS:
Locations (1):
- Swinburne University of Technology, Hawthorn, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No